CLINICAL TRIAL: NCT06366854
Title: Hemodynamic Phenotype-Based, Capillary Refill Time-Targeted Resuscitation In Early Septic Shock: The UK ANDROMEDA-SHOCK-2 Randomized Clinical Trial
Brief Title: UK ANDROMEDA-Shock-2 RCT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: Pontificia Universidad Catolica de Chile (Other); University of Rotterdam, The Netherlands (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRAS: 332418
Record Dates: First submitted 2024-04-02; First posted 2024-04-16 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): Management consists of a strategy that targets capillary refill time and individualised haemodynamic parameters, using vasopressors, fluids as guided by fluid responsiveness tests and inotropic support as guided by echocardiography.
  Interventions: Procedure: Personalised fluid and haemodynamic resuscitation
- control group (Active Comparator): Management guided by clinical team
  Interventions: Procedure: Personalised fluid and haemodynamic resuscitation

INTERVENTIONS:
Procedure: Personalised fluid and haemodynamic resuscitation — individualised resuscitation

SUMMARY:
The purpose of the trial is to test if a strategy of resuscitation guided by capillary refill time and individualised clinical hemodynamic phenotyping can improve important clinical outcomes within 28 days in septic shock patients compared to usual care.

DETAILED DESCRIPTION:
Septic shock is a life-threatening condition caused by a severe infection. It can rapidly cause multi-organ failure and is associated with a high risk of dying. Patients with septic shock need emergency treatment with intravenous fluids, antibiotics and medications to improve blood supply to all organs. However, it is clear that giving too much fluid is harmful and giving not enough fluid can make organ failure worse, too. International guidelines exist but there is still a lot of variation in how doctors apply the guideline. Further, it is likely that a "one-size-fits-all" approach does not help all patients.

Previously, the Andromeda-Shock 1 trial showed that resuscitation guided by regular monitoring of skin perfusion was associated with a lower risk of dying than resuscitation guided by regular blood tests. The UK Andromeda-Shock-2 RCT builds on this. The aim is to investigate whether an individualised approach based on monitoring of skin perfusion combined with individualised treatment of the blood pressure and circulation for 6 hours is better for patients with septic shock and reduces the risk of organ failure and dying compared to usual care.

During the study period, the investigators will also take a total of 40ml of blood and 60ml of urine for special kidney tests to evaluate kidney health and recovery of kidney function.

After the study has finished, the investigators plan to share fully anonymised results with the investigators of the international Andromeda Shock 2 trial to get as much information as possible to answer the research question and help patients in future.

ELIGIBILITY:
Inclusion Criteria:

Consecutive adult patients (≥ 18 years) with septic shock defined by Sepsis-3 consensus criteria. (ie septic shock defined as suspected or confirmed infection, hyperlactatemia and noradrenaline requirement, after a fluid load of at least 1000mL in 1 hour)

Exclusion Criteria:

Any of the following criteria preclude participation to the trial:

1. More than 4 hours since septic shock diagnosis,
2. Surgery or acute renal replacement therapy anticipated to start during the 6h intervention period
3. Active bleeding,
4. Child B-C Cirrhosis
5. Underlying disease process with a life expectancy <90 days
6. Attending clinician deems aggressive resuscitation unsuitable
7. Refractory shock (high risk of death within 24h)
8. Pregnancy
9. Concomitant severe acute respiratory distress syndrome
10. Capillary refill time cannot be accurately assessed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2027-04-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
hospital mortality | 28 days
  number of patients who died in hospital
organ support | 28 days
  time to cessation of vital organ support
length of stay | 28 days
  length of stay in hospital

SECONDARY OUTCOMES:
mortality | 60 days
  number of patients who died
vital organ support | 28 days
  number of days without vital organ support
length of stay | 60 days
  length of stay in hospital

IPD SHARING:
Plan to Share IPD: Undecided